CLINICAL TRIAL: NCT06164444
Title: Multicentre Non-inferiority Cluster Randomised Trial Testing Disposable Versus Reusable DrApes and Gowns for Green OperatiNg Theatres
Brief Title: Disposable Versus Reusable DrApes and Gowns for Green OperatiNg Theatres
Acronym: DRAGON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Christian Medical College, Vellore, India (Other); Kigali University Teaching Hospital (Other); Lagos State University (Other); Hospital Español de Mexico (Other); Christian Medical College and Hospital, Ludhiana, India (Other); Centre National Hospitalier Universitaire Hubert Koutoukou MAGA (Unknown); University for Development Studies, Tamale, Ghana (Other); Chris Hani Baragwanath Academic Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RG_22-181 - Q1085
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Surgical Site Infection
Keywords: Surgery; global surgery; SSI; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Pragmatic 1:1 international multi-centre non-inferiority cluster randomised controlled trial, with an internal pilot. Clusters are individual hospitals.
Who Masked: Outcomes Assessor
Masking Description: Patients will not specifically be blinded to the treatment allocation and those operated under non-general anaesthesia are likely to see the drapes and gowns used. However, most patients are unlikely to be able to recognise and differentiate between the different types of reusable and single use gowns and drapes, meaning unblinded patients are a low risk of bias.
  As this is a cluster randomised trial, outcome assessors are likely to know the hospital allocation and are therefore unlikely to be blinded. Assessors will receive formal training to undertake patient record review, in-person wound assessment, or telephone follow-up, as appropriate for their site. Assessors will collect detailed wound-related variables. The primary outcome of SSI will be determined by a computer-based algorithm based on the CDC criteria, using this data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Reusable drapes and gowns (Experimental): * Reusable drapes and gowns are made from cotton and polyester and are protective against fluid contamination and, to a certain extent, mechanical stress.
  * Reusable drapes and gowns are usually autoclaved and laundered using pressurised steam. This ensures that bacteria and other microorganisms are killed, sterilising the fabric so it is suitable for re-use. In this pragmatic trial, a specific sterilisation protocol is not mandated, but details of the sterilisation processes in place at each hospital will be captured in the Hospital-level Questionnaire before site opening. We may report this in a paper ahead of the main trial publication.
  Interventions: Other: Intervention: Reusable drapes and gowns
- Comparator: Disposable (single-use) drapes and gowns (Active Comparator): * Single-use surgical gowns and drapes are generally made from non-woven plastic polymers that are protective against fluid contamination and, to a certain extent, mechanical stress.
  * They are intended for use during a single operation and are then disposed of as biohazard waste for incineration.
  * Typically, four drapes are needed for an abdominal operation (two larger and two smaller drapes), although more may be needed for some procedures.
    * A range of disposable gowns are available. The choice of disposable gown will be at the hospital PI's discretion and will be captured in the Hospital-level Questionnaire.
  Interventions: Other: Comparator: Disposable (single-use) drapes and gowns

INTERVENTIONS:
Other: Intervention: Reusable drapes and gowns — Reusable drapes and gowns used during surgery.
  Arms: Intervention: Reusable drapes and gowns
Other: Comparator: Disposable (single-use) drapes and gowns — Disposable drapes and gowns used during surgery.
  Arms: Comparator: Disposable (single-use) drapes and gowns

SUMMARY:
Multicentre non-inferiority cluster randomised trial testing Disposable versus Reusable drApes and Gowns for green OperatiNg theatres. A pragmatic 1:1 international multi-centre non-inferiority cluster randomised controlled trial, with an internal pilot. Clusters are individual hospitals.

DETAILED DESCRIPTION:
Background: The World Health Organisation makes no recommendation for the use of disposable or reusable surgical drapes and gowns due to a lack of effectiveness evidence. Since disposable versions are likely to have higher financial and carbon costs, they are only justifiable if they can be proven to significantly reduce surgical site infections (SSIs).

Aim: This randomised controlled trial will assess whether reusable surgical drapes and gowns are non-inferior in reducing SSI compared to disposable drapes and gowns in patients undergoing surgery.

Design: Pragmatic 1:1 international multi-centre non-inferiority cluster randomised controlled trial, with an internal pilot. Clusters are individual hospitals.

Intervention: Reusable surgical drapes and gowns.

Comparator: Disposable (single-use) surgical drapes and gowns.

Sample size: The control group SSI event rate is estimated to be 12.5% based on previous literature. To determine whether reusable drapes and gowns are non-inferior to disposable drapes and gowns with a non-inferiority margin of 2.5% would require a total of 26,800 participants from 134 clusters, with an average of 200 participants per cluster, assuming 90% power, 2.5% one-sided alpha, intraclass correlation of 0.01 and 5% participant loss to follow up.

ELIGIBILITY:
Inclusion criteria:

* Patients with at least one incision that is ≥5cm in adults and ≥3cm in children aged under 16 years. This can include both open and minimally-invasive surgery providing at least one incision meets this criteria.
* Patients with a clean-contaminated, contaminated, or dirty surgical wound. Definitions of contamination are given in Table 2.
* Patients undergoing emergency (surgery on an unplanned admission) or elective (surgery on a planned admission) surgery.
* Any operative indication (including caesarean section).
* Patients aged 10 or over.

Exclusion criteria

* Adults with an incision <5 cm and incision <3cm in children aged under 16 years.
* Patients undergoing procedures with a clean surgical wound only.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26800 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection (SSI) | Within 30 days of surgery
  SSI according to centre for disease control (CDC) criteria:
  The infection must occur within 30-days of the index operation AND The infection must involve the skin, subcutaneous, muscular, or fascial layers of the incision AND
  The patient must have at least one of the following:
  Purulent drainage from the wound Organisms are detected from a wound swab Wound opened spontaneously or by a clinician AND, at the surgical wound, the patient has at least one of pain or tenderness; localised swelling; redness; heat; systemic fever (>38°C).
  Diagnosis of SSI by a clinician or on imaging

SECONDARY OUTCOMES:
Mortality (and likely cause) | Within 30 days of surgery
Unplanned wound opening | Within 30 days of surgery
Antibiotic prescribing for SSI | Within 30 days of surgery
Reattendance at emergency department | Within 30 days of surgery
Readmission to hospital | Within 30 days of surgery
Reoperation for SSI | Within 30 days of surgery
Total length of hospital stay | Within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Principal Investigator — University of Birmingham
Locations (1):
- CMNO, Guadalajara, Mexico

IPD SHARING:
Plan to Share IPD: No
Hospital-level data will not be released or published. Country-level analyses will only be conducted with permission of lead investigators from each participating country. Local investigators may access their data across their country to perform country-level analyses (all participating hospitals should consent to their data being used in this way).